CLINICAL TRIAL: NCT02047006
Title: Finding the Optimal Dose of Rivaroxaban in Hemodialysis Patients
Brief Title: Dose-finding of Rivaroxaban in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. An De Vriese, Head of the Department of Internal Medicine, AZ Sint-Jan AV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-Nephrology-ADV
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Renal Failure
Keywords: Hemodialysis; Rivaroxaban; AUC
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivaroxaban 10 mg (Experimental): Measurement of AUC of rivaroxaban and effect on coagulation assays:
  Rivaroxaban is given as a single oral dose of 10 mg immediately after three subsequent dialysis sessions. Patients remain in the hospital from the intake of the first dose until 48 hours after the intake of the third dose.
  Effect of dialysis on levels of rivaroxaban:
  Rivaroxaban is given as a single oral dose of 10 mg in the morning when dialysis is scheduled in the afternoon, or the previous evening when dialysis is scheduled in the morning. The interval between the two doses was at least 48 hours. Dialysis is scheduled 6 to 8 hours after the intake of rivaroxaban.
  Interventions: Drug: Rivaroxaban 10 mg

INTERVENTIONS:
Drug: Rivaroxaban 10 mg — Measurement of AUC of rivaroxaban and effect on coagulation assays:
  Venous blood samples (8.5 ml) are collected immediately before (t=0) and at t= 0,5, 1, 2, 4, 8, 12, 24, 36 and 44 hours after administration of rivaroxaban.
  Effect of dialysis on levels of rivaroxaban:
  Venous blood samples (8.5 ml) are collected at the start of dialysis (t=0) and at t=1, 2, 3 and 4 hours.

SUMMARY:
Rivaroxaban is a recently developed factor Xa (FXa) inhibitor for the prevention and treatment of thromboembolic disease. There are no data on dose adjustments in patients with severe chronic renal failure. It's use is therefore not recommended in this patient population. The present study aims to asses in 12 hemodialysis patients that require prevention of deep vein thrombosis:

1. the AUC and Cmax of 10 mg rivaroxaban
2. the effect of 10 mg rivaroxaban on coagulation assays
3. the effect of a single dialysis session on plasma levels of rivaroxaban and on anti-Xa levels
4. the safety and tolerability of rivaroxaban

DETAILED DESCRIPTION:
1. Background and Rationale:

   Vitamin K antagonists have been the standard anticoagulant treatment for decades, despite their unpredictable pharmacology and their slow onset and offset of action, requiring frequent monitoring and bridging with low molecular weight heparins (LMWH), and resulting in a substantial risk of under- and overtreatment. Patients with end-stage renal disease have an increased risk of bleeding due to their underlying disease. Therefore, anticoagulants need to be used with caution in these patients. In addition, the vitamin K antagonists are increasingly implicated in the development of vascular calcifications in this already vulnerable population. A search for alternative anticoagulants is therefore warranted.

   Rivaroxaban is a recently developed factor Xa (FXa) inhibitor for the prevention and treatment of thromboembolic disease (1). Rivaroxaban has a much lower pharmacokinetic variability and little interaction with food and drugs, contributing to consistent and predictable anticoagulation. As a consequence, routine monitoring is not required. Rivaroxaban has been shown to be effective and safe in large trials on the prevention and treatment of venous thromboembolism (2,3) and the prevention of stroke in atrial fibrillation (4).

   Rivaroxaban inhibits factor Xa in a concentration-dependent manner. Even though routine monitoring is not required, there are clinical situations in which an evaluation of its anticoagulant effect is desirable. Rivaroxaban prolongs prothrombin time (PT) and activated partial thromboplastin time (aPTTT) in a concentration-dependent manner. However, the extent of prolongation varies considerably with the type of reagent that is used. This variation cannot be reduced by conversion of PT values given in seconds to international normalized ratio values; therefore, PT and activated partial thromboplastin time are not useful for measuring the pharmacodynamic effects of rivaroxaban. Anti- Factor Xa activity is also influenced by rivaroxaban and is the most reliable method to evaluate the clinical effect of rivaroxaban (5).

   The absolute bioavailability of rivaroxaban is high (80 % - 100 %) for the 10 mg dose, with maximum plasma concentration (Cmax). appearing 2 - 4 hours after tablet intake. Intake with food does not affect rivaroxaban area under the curve (AUC) or Cmax. Rivaroxaban pharmacokinetics are approximately linear up to about 15 mg once daily. Plasma protein binding in humans is high at approximately 92 % to 95 %, with serum albumin being the main binding component. Due to the high plasma protein binding rivaroxaban is not expected to be dialysable. There are, however, no data about plasma protein binding in hemodialysis patients. Unchanged rivaroxaban is the most important compound in human plasma, with no major or active circulating metabolites being present. With a systemic clearance of about 10 l/h, rivaroxaban can be classified as a low-clearance drug. After intravenous administration of a 1 mg dose the elimination half-life is about 4.5 hours. After oral administration of a 10 mg dose the elimination becomes absorption rate limited with mean terminal half-lives of 7 to 11 hours (6,7).

   Rivaroxaban has a dual mode of elimination. Approximately 2/3 of the administered dose is metabolized to inactive metabolites in the liver, with half then being eliminated renally and the other half eliminated by the faecal route. The final 1/3 of the administered dose undergoes direct renal excretion as unchanged active substance in the urine, mainly via active renal secretion (6,7). In individuals with mild (measured creatinine clearance [CreaCl] 50-80 ml/min), moderate (CreaCl 30-49 ml/min) and severe (CreaCl 15-29 ml/min) renal impairment, rivaroxaban plasma concentrations (AUC) were increased 1.4-, 1.5- and 1.6-fold respectively, as compared with control subjects, whereas maximum plasma concentration was relatively unaffected (8). Corresponding increases in pharmacodynamic effects were more pronounced. In individuals with mild, moderate and severe renal impairment the overall inhibition of factor Xa-activity was increased by a factor of 1.5, 1.9 and 2.0 respectively, as compared to healthy volunteers; prolongation of PT was similarly increased by a factor of 1.3, 2.2 and 2.4 respectively (8). There are no data in patients with CreaCl < 15 ml/min. Based on these data, dosing guidelines for patients with renal failure have been issued. No dose adjustment is necessary in patients with mild renal impairment (CreaCl 50-80 ml/min) or moderate renal impairment (CreaCl 30-49 ml/min). In patients with severe renal impairment (CreaCl 15-29 ml/min), rivaroxaban is to be used with caution. Use is not recommended in patients with CreaCl < 15 ml/min (6,7).
2. Study design A two-centre, non-blinded cohort study.
3. Study objectives 1) To measure the AUC and Cmax of 10 mg rivaroxaban in hemodialysis patients 2) To assess the effect of 10 mg rivaroxaban on coagulation assays in hemodialysis patients:

   * anti-Xa assay
   * prothrombin assay 3) To assess the effect of a single dialysis session on plasma levels of rivaroxaban and on anti-Xa levels 4) To assess safety and tolerability of rivaroxaban in hemodialysis patients
4. Study subjects

   1. Enrolment procedure The study protocol will be discussed with eligible patients. All patients under treatment in the participating centers that meet the in- and exclusion criteria that give informed consent will be included.
   2. Planned number of participants 12 patients
   3. Inclusion criteria

      * age ≥18 year
      * signed informed consent
      * chronic hemodialysis patients without immediate life-threatening conditions, dialysed three times a week for at least three months
      * requiring anticoagulation for the prevention of deep venous thrombosis
   4. Exclusion criteria

      * residual renal function, as defined by a residual diuresis of >50 ml/day
      * known intestinal malabsorption
      * inability to take oral medication
      * mechanical heart valve
      * inability to stop co-medication that causes major interactions with rivaroxaban (e.g. ketoconazole, itraconazole, voriconazole, posaconazole, ritonavir)
      * severe liver dysfunction Child-Pugh grade C

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 year
* signed informed consent
* chronic hemodialysis patients without immediate life-threatening conditions, dialysed three times a week for at least three months
* requiring anticoagulation for the prevention of deep venous thrombosis

Exclusion Criteria:

* residual renal function, as defined by a residual diuresis of >50 ml/day
* known intestinal malabsorption
* inability to take oral medication
* mechanical heart valve
* inability to stop co-medication that causes major interactions with rivaroxaban (e.g. ketoconazole, itraconazole, voriconazole, posaconazole, ritonavir)
* severe liver dysfunction Child-Pugh grade C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics and pharmacodynamics of rivaroxaban in hemodialysis patients | AUC for 48 hours
  1. To measure the AUC and Cmax of 10 mg rivaroxaban in hemodialysis patients
  2. To assess the effect of 10 mg rivaroxaban on coagulation assays in hemodialysis patients:
     * anti-Xa assay
     * prothrombin assay

SECONDARY OUTCOMES:
Dialytic removal of rivaroxaban | 4 hours
  To assess the effect of a single dialysis session on plasma levels of rivaroxaban and on anti-Xa levels
Safety and tolerability of rivaroxaban in hemodialysis patients | 2 weeks
  Subjective tolerability is evaluated by questioning the patients about any adverse events or by spontaneous reporting of adverse events. Objective tolerability is evaluated by monitoring vital signs and routine clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: An S De Vriese, MD, PhD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (2):
- Belgium (2):
  - OLV Aalst, Aalst
  - AZ Sint-Jan Brugge-Oostende AV, Bruges